CLINICAL TRIAL: NCT06139367
Title: A Randomized, Open, Parallel, Single Center Phase I Clinical Trial to Evaluate the Effect of Food on the Pharmacokinetics of TQB3454 Tablets in Healthy Adult Subjects.
Brief Title: A Clinical Trial of TQB3454 Tablets in Healthy Adult Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TQB3454-I-03
Record Dates: First submitted 2023-11-15; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Biliary Carcinoma
Keywords: Food effect

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TQB3454 tablets under fast condition (Experimental): TQB3454 tablets 600mg, take one dose orally under fast condition.
  Interventions: Drug: TQB3454 tablets
- TQB3454 tablets under fed condition (Experimental): TQB3454 tablets 600mg, take one dose orally under fed condition.
  Interventions: Drug: TQB3454 tablets

INTERVENTIONS:
Drug: TQB3454 tablets — TQB3454 is a Isocitrate dehydrogenase 1 (IDH1) mutation inhibitor.

SUMMARY:
This is a randomized, open, parallel, single center phase I clinical trial to evaluate the impact of food on the pharmacokinetics of TQB3454 tablets in healthy adult subjects. The aim is to evaluate the impact of food on the pharmacokinetics as well as the safety after single dose of TQB3454 tablets taken orally by Chinese healthy adult subjects, with pharmacokinetic indicators as the primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Sign an informed consent form before the experiment and fully understand the content, process, and potential adverse reactions of the study;
* Able to complete the study according to the requirements of the protocol;
* Subjects aged 18-65 (inclusive);
* Body mass index (BMI) ≥ 18 and ≤ 28 kg/m^2, and male's weight ≥ 50 kg and female's weight ≥ 45 kg;
* Health status: No mental abnormalities, no history of severe neurological, respiratory, digestive, urinary, endocrine, and metabolic abnormalities;
* The subjects have no pregnancy plan, voluntarily take effective contraceptive measures, and no plans to donate sperm or eggs, from the date of signing the inform consent (14 days before signing the inform consent for female subjects) to at least 6 months after the last administration.

Exclusion Criteria:

* Subjects with allergic constitution or a history of allergies to two or more foods or drugs;
* Subjects who have experienced arterial/venous thrombosis events within 6 months, such as cerebrovascular accidents (including temporary ischemic attacks), deep vein thrombosis, and pulmonary embolism;
* Suffering from ≥ Level 2 myocardial ischemia or infarction, arrhythmia (including QTc ≥ 450 ms for male, QTc ≥ 470 ms for female), and ≥ Level 2 congestive heart failure (New York Heart Association (NYHA) classification);
* Those with multiple factors that affect oral medication (such as inability to swallow, gastrointestinal diseases);
* Have taken any prescription, over-the-counter, vitamin product, or herbal medicine within one month before the first administration;
* Take CYP3A4 inhibitors or inducers within one month before the first administration or before the study medication;
* Those who have taken a special diet (including grapefruit, etc.) or engaged in vigorous exercise within 14 days before the first administration or have other factors that affect drug absorption, distribution, metabolism, excretion, etc.;
* Abnormal and clinically significant physical examination, vital signs, electrocardiogram, and laboratory tests during the screening period;
* Donated blood or experienced significant blood loss (>450 mL) within 3 months prior to taking the study drug;
* Participated in any clinical trial and took any investigational drug within 3 months prior to taking the study drug;
* Smoke at least 5 cigarettes per day within 3 months prior to the study;
* Positive alcohol breath test or history of alcoholism within 2 weeks prior to screening (drinking 14 units of alcohol per week: 1 unit=360 mL of beer or 45 mL of 40% alcohol or 150 mL of wine);
* Drug screening positive or those who have used drugs in the past 3 months prior to the study;
* Inability to tolerate venous puncture for blood collection or poor vascular condition;
* The subject is unable to complete the experiment due to personal reasons;
* Other conditions that it is considered not suitable for enrollment assessed by the investigators.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Peak concentration (Cmax) | pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 264, 330 hours after dose.
  Maximum plasma drug concentration
Area under the time-concentration curve from 0 to t hours (AUC0-t) | pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 264, 330 hours after dose.
  Area under the plasma concentration-time curve from the time of first dose to the time of the last measurable concentration.
Area under the time-concentration curve from 0 to infinity (AUC0-∞) | pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 264, 330 hours after dose.
  Area under the plasma concentration-time curve from the time of first dose extrapolated to infinity
Time to peak (Tmax) | pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 264, 330 hours after dose.
  Time to reach maximum plasma concentration after drug administration
Elimination half-life (t1/2) | pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 264, 330 hours after dose.
  The time it takes for the blood concentration of a drug to decrease from its highest value to half in the body.
Apparent volume of distribution (Vd/F) | pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 264, 330 hours after dose.
  The ratio of the amount of drug in the body to the concentration in the blood.
Apparent clearance (CL/F) | pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 264, 330 hours after dose.
  Apparent total clearance of the drug from plasma after oral administration.
Elimination rate constant (λz) | pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 264, 330 hours after dose.
  Terminal disposition rate constant/terminal rate constant
Lag time (tlag) | pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 264, 330 hours after dose.
  The time required from the start of administration to the appearance of the drug in the blood.
Percentage of residual area (AUC% Extrap) | pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 264, 330 hours after dose.
  Residual area as a percentage of the entire area under curve.

SECONDARY OUTCOMES:
Adverse event rate | Before the first administration to 360 hours after the last administration.
  The incidence of adverse events (AEs), abnormal laboratory test values, and severe adverse events (SAEs).
Adverse event severity | Before the first administration to 360 hours after the last administration.
  The severity of adverse events (AEs), abnormal laboratory test values, and severe adverse events (SAEs).

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Qingdao University, Qingdao, Shandong, China